CLINICAL TRIAL: NCT00216554
Title: A Multicenter, Open-Label Study to Evaluate Safety and Efficacy of Risperidone as Adjunctive Therapy to Mood Stabilizers in the Long-term Treatment of Bipolar Mania
Brief Title: The Safety and Efficacy of Risperidone as Adjunctive Therapy to Mood Stabilizers in the Long-term Treatment of Bipolar Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005068
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; risperidone; Adjunctive therapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to evaluate effect of risperidone as a long-term combination therapy to mood stabilizers in the treatment of bipolar mania

DETAILED DESCRIPTION:
The use of mood stabilizers such as lithium and carbamazepine is known to be effective for preventing and treating bipolar disorder. But the use of antipsychotic drugs is more effective in patients suffering severe episodes of mania as it elicits behavioral changes and spurs the effects of mood stabilizers. Antipsychotic drugs are used for patients who failed to respond to mood stabilizers or for the acute management of manic episodes associated with bipolar disorders.

This study aims to evaluate the safety and efficacy of risperidone as an adjunctive therapy to mood stabilizers in the long-term treatment (6months) of bipolar disorder using various assessment instruments, including the Young Mania Rating Scale. The Simpson-Angus Rating Scale will be also employed to assess the presence of extrapyramidal side effects and other adverse events. The patients will receive orally 0.5, 1, 2 mg risperidone tablet once daily for 6 months

ELIGIBILITY:
Inclusion Criteria:

* In- or out-patient
* Diagnosis of bipolar I disorder
* most recent episode manic with or without psychotic features
* YMRS > 20 (manic)
* Need antipsychotic combination on the basis of clinicians' experience

Exclusion Criteria:

* Rapid cycling
* Risk of suicide or violence
* History of Substance dependence within 3 months
* Comorbidities
* Unstable medical illness
* Previous sensitivity history to risperidone
* Pregnant woman or those without proper contraception
* History of clozapine and one cycle of depot use prior to entry
* History of treatment resistance: at least two mood stabilizers
* Prior history of active treatment with risperidone
* As for patients having wash-out period, patients that show 25% or more decrease in YMRS at baseline as compared to that at enrollment time, should be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2004-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The change in YMRS score from baseline at 6 months

SECONDARY OUTCOMES:
The change from baseline in Clinical Global Impression-Severity (CGI-S) score at 6 months; The change from baseline in HAMD score at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.